CLINICAL TRIAL: NCT00356681
Title: A Randomized Phase 2 Trial of Double-Blind, Placebo Controlled AMG 706 in Combination With Paclitaxel, or Open-Label Bevacizumab in Combination With Paclitaxel, as First Line Therapy in Women With HER2 Negative Locally Recurrent or Metastatic Breast Cancer
Brief Title: A Study of AMG 706 or Bevacizumab, in Combination With Paclitaxel Chemotherapy, as Treatment for Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to close study
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20050225; CIRG/TORI 010
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-09

CONDITIONS: Breast Neoplasms; Breast Tumors; Breast Cancer; Locally Recurrent and Metastatic Breast Cancer
Keywords: AMG 706; Paclitaxel; Metastatic Breast Cancer; Antiangiogenic; Bevacizumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; motesanib diphosphate; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A Placebo (Placebo Comparator): Blinded AMG 706 placebo plus paclitaxel
  Interventions: Drug: AMG 706 placebo; Drug: Paclitaxel
- Arm B Experimental (Experimental): Blinded AMG 706 plus paclitaxel
  Interventions: Drug: AMG 706; Drug: Paclitaxel
- Arm C Comparator (Active Comparator): Open-label bevacizumab plus paclitaxel
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: AMG 706 placebo — Blinded placebo
  Arms: Arm A Placebo
Drug: Bevacizumab — Bevacizumab is a recombinant, humanized anti-VEGF monoclonal antibody.
  Other Names: Avastin
  Arms: Arm C Comparator
Drug: AMG 706 — AMG 706 is a small organic molecule that has been shown in preclinical pharmacology and PK studies to be a potent, oral, multi-kinase inhibitor with anti-angiogenic and anti-tumor activity achieved by selectively targeting all known VEGF, PDGF and Kit receptors.
  Other Names: motesanib diphosphate
  Arms: Arm B Experimental
Drug: Paclitaxel — Paclitaxel is an antineoplastic agent that acts by promoting and stabilizing the polymerization of microtubules.

SUMMARY:
To determine if treatment with paclitaxel plus AMG 706 is superior to paclitaxel plus AMG 706 placebo in subjects with HER2 negative locally recurrent or metastatic breast cancer. Also to estimate differences between treatment with paclitaxel plus AMG 706 and paclitaxel plus bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast with locally recurrent or metastatic disease.
* Measurable disease by RECIST guidelines.
* Tumor (primary or metastatic) must be HER2 negative.
* Adequate organ and hematologic function. Exclusion:
* Taxane treatment within 12 months prior to registration.
* Prior chemotherapy for locally recurrent or metastatic breast cancer (prior endocrine therapy is permitted).
* Prior radiation therapy, radiofrequency ablation, percutaneous cryotherapy or hepatic chemoembolization on all sites of measurable disease.
* Current or prior history of central nervous system metastases.
* Peripheral neuropathy ≥ grade 2 (CTCAE v3.0) at registration.
* History of arterial or venous thrombosis within 1 year prior to registration.
* History of bleeding diathesis or bleeding within 14 days of registration.
* Uncontrolled hypertension (systolic >145 mmHg; diastolic >85 mmHg).
* Clinically significant cardiac disease within 12 months of registration.
* Known HIV positive, hepatitis C positive or hepatitis B surface antigen positive.
* Prior treatment with VEGFr targeted therapies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2006-12; Primary Completion 2009-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Objective response rate, measured radiologically and assessed by an independent review committee. | Last patient enrolled + 16 weeks of treatment

SECONDARY OUTCOMES:
Progression free survival, duration of response, clinical benefit rate (percentage of subjects with complete response, partial response or stable disease lasting >24 weeks), overall survival and incidence of adverse events. | >24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Martin M, Roche H, Pinter T, Crown J, Kennedy MJ, Provencher L, Priou F, Eiermann W, Adrover E, Lang I, Ramos M, Latreille J, Jagiello-Gruszfeld A, Pienkowski T, Alba E, Snyder R, Almel S, Rolski J, Munoz M, Moroose R, Hurvitz S, Banos A, Adewoye H, Hei YJ, Lindsay MA, Rupin M, Cabaribere D, Lemmerick Y, Mackey JR; TRIO 010 investigators. Motesanib, or open-label bevacizumab, in combination with paclitaxel, as first-line treatment for HER2-negative locally recurrent or metastatic breast cancer: a phase 2, randomised, double-blind, placebo-controlled study. Lancet Oncol. 2011 Apr;12(4):369-76. doi: 10.1016/S1470-2045(11)70037-7. Epub 2011 Mar 21. PMID 21429799
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com